CLINICAL TRIAL: NCT04966520
Title: Repetitive Intermittent Accelerated Theta-burst Transcranial Stimulation(iTBS) as a Potential Intervention for Chemotherapy Induced Cognitive Deficits (CICD)- a Pilot Clinical Trial to Explore Feasibility and Efficacy
Brief Title: Accelerated Neuromodulation to Alleviate Cognitive Deficits Due to Cancer Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sneha Phadke (Other)
Collaborators: American Cancer Society-Holden Comprehensive Cancer Society (Unknown); Fraternal Order of Eagles (Iowa) (Unknown)
Responsible Party: Sponsor-Investigator, Sneha Phadke, Clinical Associate Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202101546
Record Dates: First submitted 2021-06-10; First posted 2021-07-19 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Cancer
Keywords: neuromodulation; chemo-brain
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Accelerated repetitive intermittent theta-burst transcranial stimulation (iTBS) or sham (Experimental): Patients will participate in the prospective longitudinal research protocol over a period of 1.5 months.
  Treatment will include 8 visits of either accelerated repetitive intermittent theta-burst transcranial stimulation (iTBS) or iTBS sham stimulation. Patients will be informed that iTBS sham stimulations will be part of the protocol (but will be blind to when treatment/sham will be administered).
  Interventions: Other: Accelerated repetitive intermittent theta-burst transcranial stimulation (iTBS)

INTERVENTIONS:
Other: Accelerated repetitive intermittent theta-burst transcranial stimulation (iTBS) — Accelerated iTBS will be used to stimulate the regions of interest of mPFC and L-DLPFC nodes in cancer survivors or patients.
  Accelerated iTBS will be administered in a single half-day period to allow for a 50minutes interval between any two treatments to minimize interference effects between treatments. Thus, there will be ~10 minute sessions of stimulation x 2 applications per node x 2 nodes (L-DLPFC, mPFC) = 40 total minutes of daily stimulation - each session delivers 1800 pulses in a 5 Hz triplet burst frequency, 2 second trains with intertrain interval of 8 seconds; triplets occur with 50 Hz frequency, as per standard iTBS protocols for depression treatment. The treatment will be offered for five consecutive days.

SUMMARY:
This project is aimed at the discovery of neuro-modulation techniques that may alleviate chemotherapy induced cognitive deficits (CICD), especially in executive (higher-order) cognitive function (EF).

DETAILED DESCRIPTION:
The specific aim for this study is to use magnetic resonance spectroscopy (MRS), self-report, and neuropsychological testing to identify changes in brain metabolite concentrations/ratios and changes in EF deficits associated with chemotherapy, before and after accelerated theta-burst transcranial stimulation (iTBS). The secondary aim is to assess for any association of changes in executive function with brain metabolite concentrations.

ELIGIBILITY:
Inclusion Criteria:

* Women or men with a history of non-metastatic cancer who have completed definitive curative cancer therapy
* Received cytotoxic chemotherapy as a part of their therapy for cancer and at least one month has passed since the final cytotoxic chemotherapy treatment
* ≥ 18 years of age at time of cancer diagnosis and receipt of chemotherapy
* Patients must report subjective symptoms of "chemo-brain" (memory loss, difficulty with concentration, word-finding difficulties) with a FACT-Cog perceived cognitive impairment score < 60
* Ability to sign informed consent and comply with study procedures

Exclusion Criteria:

* Patients with a recurrence of cancer or those with current metastatic disease
* Patients with a history or current diagnosis of brain metastasis
* Patients with a history or current diagnosis of a primary brain tumor
* Patients with a history of brain surgery or brain radiation
* Patients receiving maintenance systemic therapy for cancer, other than endocrine therapy
* Patients who cannot produce or request adequate medical record documentation to ensure they meet inclusion and exclusion criteria
* Women who are currently pregnant
* History of childhood cancer or receipt of chemotherapy in childhood (<age 18). Developmental insult to the PFC, can be associated with long-term, durable and sometime debilitating cognitive deficits. Hence, we avoid any cognitive confounds that maybe related to this issue.
* Patients with a weight over 250 lbs., as these patients would not fit in the MRI scanner used in the protocol
* Patients who require benzodiazepines for MRI due to claustrophobic anxiety
* Patients with chest wall tissue expanders or other retained 7 Tesla MRI-incompatible metal. Any other specific contraindication to TMS or MRI not already listed above, including:
* (a) any implanted device in the head, neck or upper body (e.g. cochlear implant, cranial or other electrodes, pacemaker or defibrillator, medication pump, stent, aneurysm clip, etc.)
* (b) personal history of seizures or epilepsy, personal history of multiple concussions or unexplained loss of consciousness. This will be determined by physician judgement
* History of adverse reaction to previous TMS or MRI exposure
* Active substance use disorder in the past 6 months, excluding tobacco use disorder, as diagnosed by study physicians

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-07-18 (Actual); Study Completion 2023-07-18 (Actual)

PRIMARY OUTCOMES:
Mean changes in executive cognitive function between pre and post application of iTBS treatment protocol | 1.5 months
  Executive cognitive function will be quantified using technician administered Color Word Interference Test, Category Fluency, Tower of Hanoi, Card Sort and Strategy Application Task (Shallice &Burgess) tests, and the self-report Functional Assessment of Cancer Therapy - Cognitive Scale (FACT-COG) (Dyk et al.). Executive Function (EF) is measured by utilizing standardized test scores adapted from the Delis-Kaplan Executive Function Scales (D-KEFS battery) (Homack et al.). FACT-COG, Category Fluency and Strategy Application Task use raw scores. All EF measures used in this battery form a part of a normative database created and maintained by the principle investigator of this study. An overall score of EF is computed by averaging the Z scores of each test. Higher score on each test represents better performance.
Mean changes in brain metabolite concentrations between pre and post application of iTBS treatment protocol | 1.5 months
  Proton Magnetic Resonance Spectroscopy will be used to quantify brain metabolite concentrations in parts per million. Brain metabolites under evaluation include: glutamine, glutamate, N-acetyl aspartate, choline, and creatine.

CONTACTS AND LOCATIONS:
Overall Officials: Sneha Phadke, DO, Principal Investigator — University of Iowa Hospitals & Clinics
Locations (1):
- University of Iowa Hospitals & Clinics, Iowa City, Iowa, United States